CLINICAL TRIAL: NCT06801158
Title: Adverse Drug Reactions to Cancer Therapies in Patients with Depression: Insights from VigiBase
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: Pharmacol20241101
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Adverse Effects of Medical Drugs
Keywords: adverse effects; oncology; vigibase
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Patients with an adverse effect of interest (or with a severity criteria of that AE)
  Interventions: Drug: use of anticancer drugs in monotherapy or in combination therapy
- Patients without an adverse effect of interest (or without a severity criteria of that AE)
  Interventions: Drug: use of anticancer drugs in monotherapy or in combination therapy

INTERVENTIONS:
Drug: use of anticancer drugs in monotherapy or in combination therapy — ICSRs involving antineoplastic or immunomodulating agents were included.

SUMMARY:
Importance:

Depression is prevalent among oncology patients and may influence the perception, reporting, and severity of adverse events (AEs) related to cancer therapies. Understanding this association is crucial for optimizing treatment outcomes and improving patient quality of life.

Objective:

To evaluate the association between depression and the reporting and severity of AEs among oncology patients using data from VigiBase®, the World Health Organization's global pharmacovigilance database.

Design:

This pharmacovigilance study employed a case/non-case disproportionality analysis using Individual Case Safety Reports (ICSRs) from 1968 to 2024. Multivariable analyses were conducted to adjust for potential confounders, such as age and sex.

Setting:

The study utilized data from VigiBase®, a global pharmacovigilance database containing reports from over 120 countries.

Participants:

ICSRs involving antineoplastic or immunomodulating agents were included. Depression was identified through antidepressant use, yielding 428,102 reports for patients on antidepressants and 8,376,761 for those not on antidepressants.

Exposure:

Oncology patients receiving antidepressant therapy were compared to those not receiving such treatment.

Main Outcome and Measures:

The primary outcome was the reporting of serious AEs (e.g., hospitalization, life-threatening events). Secondary outcomes included the 20 most frequently reported AEs among oncology patients, with comparisons made between those treated with and without antidepressants.

ELIGIBILITY:
Inclusion Criteria:

* ICSRs were limited to those involving liable antineoplastic or immunomodulating agents (per the Anatomical Therapeutic Chemical (ATC) Classification code L; hereafter referred to as antineoplastics)

Exclusion Criteria:

* Suspect of duplication

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Antidepressants were employed as a proxy for identifying patients experiencing depression. These agents were identified according to the ATC classification for antidepressants (code N06A).
Sampling Method: Probability Sample
Enrollment: 8804863 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-16 (Actual)

PRIMARY OUTCOMES:
reporting of serious AEs | 1964 to 2024

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No
Data belong to the WHO Uppsala Monitoring Center